CLINICAL TRIAL: NCT00319059
Title: The Influence of the 34C>T Variant in the AMPD1 Gene on Individual Susceptibility for Ischemia-reperfusion.
Brief Title: The Influence of the 34C>T Variant in the AMPD1 Gene Ischemic Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AMPD-Annexin
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: AMPD; Ischemic Tolerance

INTERVENTIONS:
Drug: systemic administration of 99mTc-HYNIC-Annexin A5
Behavioral: 10 minutes of ischemic handgripping

SUMMARY:
Previous epidemiological studies have shown that in cardiovascular patients, the 34C>T variant in the gene encoding for the enzyme Adenosine Mono Phosphate Deaminase (AMPD1) is associated with prolonged survival.

The 34 C>T variant encodes a severely truncated, metabolically inactive protein. We hypothesize that during ischemia, in these patients AMP in preferentially converted into adenosine instead of IMP. Adenosine receptor stimulation, in turn, will increase resistance to ischemia-reperfusion in the myocardial tissue.

To test this hypothesis, 7 male healthy volunteers heterozygous for the 34C>T variant will be selected from 100 healthy volunteers, which we have previously genotyped. These subjects will be compared with 7 matched control subjects. Individual ischemic tolerance will be assessed in the thenar muscle using 99mTc-Annexin A5 scintigraphy.

Briefly, the circulation of the nondominant forearm will be interrupted for 10 minutes by inflation of an upperarm cuff to 200mmHg en concomitantly, the subjects will perform isometric rhythmic handgripping until exhaustion. Immediately upon reperfusion, 400 MBq of 99mTc-Annexin A5 will be administered intravenously. Finally, 1 and 4 hours post-injection, scintigrapghi imaging of both hand will be performed. Targeting of annexin A5 will be expressed as percentage difference between the experimental and control hand.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-40 years
* healthy
* AMPD1 34C>T variant (heterozygous) or matched control

Exclusion Criteria:

* cardiovascular / pulmonary disease
* diabetes / hypertension

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2006-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
99mTc-Annexin A5 targeting

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, PhD, Principal Investigator — Radboud University Medical Center